CLINICAL TRIAL: NCT06721611
Title: A Comprehensive Optical Blood Pressure Assessment Tool to Identify Cases of Unscreened Hypertension Across an Active Population in the U.S.: a Prospective Single-center Observational Clinical Study.
Brief Title: A Comprehensive Optical Blood Pressure Assessment Tool to Identify Cases of Unscreened Hypertension Across an Active Population in the U.S.
Acronym: CATCH-US
Status: Withdrawn | Type: Observational
Why Stopped: The study was aborted by the sponsor.
Sponsor: Nucor (Industry)
Responsible Party: Sponsor
Other Study IDs: CATCH-US
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CATCH-US cohort: Non-hypertensive Nucor employees that accept to receive and wear continuously for 28 days an optical blood pressure monitoring device (Aktiia 24/7 device)
  Interventions: Device: Optical Blood Pressure Monitoring Device (Aktiia G1)

INTERVENTIONS:
Device: Optical Blood Pressure Monitoring Device (Aktiia G1) — Non-hypertensive Nucor employees that accept to wear an optical blood pressure monitoring device (Aktiia 24/7 device) to screen for and identify potential undiagnosed hypertension.
  100 participants. Each participant will wear the device continuously for 28 days.

SUMMARY:
To screen for and identify subjects with potential undiagnosed hypertension using an optical blood pressure monitoring device across an active workforce population in the US (Nucor employees).

DETAILED DESCRIPTION:
100 voluntary Nucor facility employees with no previous diagnosis of hypertension will be recruited and will receive an optical blood pressure monitoring device (Aktiia G1 Device) that is a miniature bracelet placed in the wrist and measure blood pressure continuously without inflating.

Each participant will wear the device continually during 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 25 to 70 years old.
2. People who self-report that they do not have a diagnosis of hypertension.
3. People employed as a Nucor team member.
4. People who can read and speak English.
5. People who use either an iOS or Android smart phone.
6. Subjects who agree to follow study procedures.
7. Subjects who have signed the informed consent form.

Exclusion Criteria:

1. Subjects with a known diagnosis of i. atrial fibrillation ii. congestive heart failure iii. heart valve disease iv. pheochromocytoma v. Raynaud's disease vi. arm lymphedema.
2. Subjects who take insulin.
3. Subjects who are on hemodialysis.
4. Women who are known to be pregnant.
5. Subjects whose arms shake uncontrollably or are paralyzed (cannot move).
6. Subjects who do not have two arms.
7. Subjects with upper arm circumference < 22cm or > 42cm.
8. Subjects with wrist circumference > 23cm.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 subjects aged 25 to 70 years old who do not have a known diagnosis of hypertension and are employed at the Nucor Corp facility.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-07-16 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects with undiagnosed hypertension | Each participant will wear the device continuously for 28 days.
  Analysis of the percentage of subjects with undiagnosed hypertension defined as an average daytime SBP>130 or DBP>80 mmHg over the initial 7 days of the Aktiia 24/7 device use.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucor, Charlotte, North Carolina, United States